CLINICAL TRIAL: NCT02049840
Title: The European Study of Altis Single Incision Sling System for Female Stress Urinary Incontinence
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU016
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Female sling; Stress Urinary Incontinence; Urination Disorders; Urologic Diseases
MeSH Terms: conditions — Urinary Incontinence, Stress; Urination Disorders; Urologic Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, post-market, single arm, mutlicenter
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altis Single Incision Sling System (Experimental): Altis Single Incision Sling System
  Interventions: Device: Altis Single Incision Sling System

INTERVENTIONS:
Device: Altis Single Incision Sling System — Altis Single Incision Sling (SIS) System is a permanently implantable synthetic sling for the surgical treatment of Stress Urinary Incontinence

SUMMARY:
This is a prospective, post-market, single arm, multicenter study comparing Baseline data to the 12 month and 36 month data in 136 female patients with Stress Urinary Incontinence

DETAILED DESCRIPTION:
This study is a prospective, European Post-Market, one non-controlled arm, multi-centre clinical trial conducted at up to 10 centers in Europe. It is designed to get more clinical information for users (uro-gynecologists) of the Altis Single Incision Sling System for female stress urinary incontinence treatment in terms of objective and subjective cure rate, quality of life improvement, patient satisfaction and safety, especially in long term follow-up (3 years). Clinical data will be collected at baseline, implantation procedure, post-operative at 6 weeks, 6 months, 1, 2 and 3 years

ELIGIBILITY:
Inclusion Criteria:

* The subject is female at least 18 years of age
* The subject uses a method of contraception considered effective by the investigator or is not of child-bearing potential
* The subject is able and willing to complete all procedures and follow-up visits indicated in this protocol.
* The subject has confirmed stress urinary incontinence (SUI) through cough stress test at baseline.
* The subject has failed first line treatments (non-invasive therapies, eg. behavioral modification, Pelvic Floor/Kegel exercises, or biofeedback) with good compliance for the treatment

Exclusion Criteria:

* The subject had a prior surgical SUI treatment (including bulking agent).
* The subject is having a concomitant Pelvic Organ Prolapse repair or hysterectomy during Altis procedure.
* The subject has incontinence due to neurogenic causes (e.g. multiple sclerosis, spinal cord/brain injury, cerebrovascular accident, detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions).
* The subject has predominant or uncontrolled or primary urge incontinence according to investigator judgment
* The patient has detrusor overactivity determined through urodynamics
* The subject has intrinsic sphincter deficiency defined urodynamically as a Maximal Urethral Closure Pressure < 20 cm H2O and/or Valsalva Leak Point Pressure < 60 cm H2O
* The subject has atonic bladder, a persistent post void residual (PVR) > 100 ml or chronic urinary retention.
* The subject has untreated urinary malignancy
* The subject has undergone radiation or brachy therapy or chemotherapy to treat pelvic cancer.
* The subject has urethrovaginal fistula or urethral diverticulum or congenital urinary anomalies
* The subject has serious bleeding disorder or requires anticoagulant therapy
* The subject is pregnant and/or is planning to get pregnant in the future.
* The subject has a Body Mass Index ≥ 35 (obese class II).
* The subject has a contraindication to the surgical procedure according to the the Altis SIS System IFU.
* The subject has an active urogenital infection or active skin infection in region of surgery mainly at the time of implantation.
* The subject is enrolled in a concomitant clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who meet the criteria of cure at 12 months | 1 year
  Cure is defined as negative Cough Stress Test (CST) and an answer "no" to question 3 "Do you usually experience urine leakage related to coughing, sneezing, or laughing?" of the UDI-6 questionnaire

SECONDARY OUTCOMES:
Proportion of subjects who have a negative cough stress test at each visit | 6 weeks, 6 months, 1 year, 2 year, 3 year
Proportion of subjects who meet the criteria of cure at each other visit | 6 weeks, 6 months, 2 year, 3 year
  Cure is defined as negative Cough Stress Test (CST) and an answer "no" to question 3 "Do you usually experience urine leakage related to coughing, sneezing, or laughing?" of the UDI-6 questionnaire
Subject continence status measured by the 24-hour pad weight | 6 weeks, 1 year
  The continence status will be described : Proportion of subjects who meet the criteria of dryness defined as a pad weight of less than 8 grams for the current practice Proportion of subjects who meet the criteria of improvement defined as at least a 50% reduction in pad weight from baseline
Assessment of self reported symptoms and subject QoL through the scoring of validated questionnaires: ICIQ-UI SF, I-QOL, UDI-6 and IIQ-7 | 6 weeks, 6 months, 1 year, 2 year, 3 year
  The scores of ICIQ-UI short form, I-QOL, UDI-6 and IIQ-7 will be describe at each visit as continuous variables. The evolution of scores from baseline will be presented
Postoperatively subject impression of improvement (via PGI-I questionnaire) and satisfaction at each post-operative visit | 6 weeks, 6 months, 1 year, 2 year, 3 year
Assessment of Qmax variations | 6 weeks, 1year
  Qmax (maximum flow rate in uroflowmetry section) raw value (at baseline, 6 weeks and 12 months) and absolute and relative variations from baseline et 6 weeks and 12 months will be described
Assessment of PVR variations | 6 weeks, 1 year
  PVR (Post void residual urine volume) raw value (at baseline, 6 weeks and 12 months) and absolute and relative variations from baseline et 6 weeks and 12 months will be described
Assessment of the operation duration and the type of anaesthesia used | Operative period
Assessment of device and procedure related adverse events | Operative period, 6 weeks, 6 months, 1 year, 2 year, 3 year
  All device or procedure related Adverse Events (AE) will be summarized and reported as the number and percentage of subjects having this AE and as the number and percentage of AE in Safety population.
Assessment of postoperative pain | operative period, 6 weeks, 6 months, 1 year
  Visual Analogue Scale from 0 "no pain" to 10 "extreme pain"

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Cornu, Pr, Principal Investigator — Centre Hospitalier Universitaire de Rouen - Hôpital Charles Nicolle
Locations (13):
- France (6):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital de la Conception, Marseille
  - Centre Hospitalier Universitaire Carémeau - Gyneacology, Nîmes
  - Centre Hospitalier Universitaire Carémeau, Nîmes
  - Centre Hospitalier Universitaire de Rouen - Hôpital Charles Nicolle, Rouen
  - Nouvel Hôpital Civil, Strasbourg
- Germany (2):
  - Isarklinikum, München
  - Chirurgische Klinik München - Bogenhausen GmbH, München
- Ospedale Garibaldi-Nesima, Catania, Italy
- Isala Klinieken Locatie Sophia, Zwolle, Netherlands
- Spain (3):
  - Hospital Universitario La Ribera, Alzira, Valencia
  - Hospital de Sagunto, Sagunto, Valencia
  - Fundacion Jimenez Diaz, Madrid